CLINICAL TRIAL: NCT04936841
Title: Phase II Study of Bempegaldesleukin (NKTR-214) Together With Palliative Radiation and Anti-PD-1 Checkpoint Blockade in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Bempegaldesleukin (NKTR-214) With Radiation and Anti-PD-1 Immunotherapy for Head and Neck Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study closed by the sponsor
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW20092; A533300 (Other: UW Madison); SMPH/HUMAN ONCOLOGY (Other: UW Madison); Protocol Version 4/19/2021 (Other: UW Madison); 2021-0141 (Other: Health Science IRB)
Record Dates: First submitted 2021-06-10; First posted 2021-06-23 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — bempegaldesleukin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NKTR-214, anti-PD therapy plus Palliative Radiation (Experimental): Cycle 1 consists of anti-PD-1 therapy (200mg) and NKTR-214 (0.006 mg/kg3 administered intravenously), followed by palliative radiation (8 Gy x 3 or 4 Gy x 5 fractions) combined with anti-PD-1 therapy and NKTR-214 in cycle 2.
  In subsequent cycles participants will receive NKTR-214 and anti-PD-1.
  Interventions: Drug: NKTR-214; Drug: anti-PD-1 therapy; Radiation: Palliative Radiation

INTERVENTIONS:
Drug: NKTR-214 — Bempegaldesleukin (NKTR-214) is an immunotherapeutic protein prodrug specifically designed to activate the patient's immune system for the treatment of cancer by providing a controlled, sustained signal to the interleukin-2 (IL-2) receptor pathway (pharmacological classification: immunostimulatory interleukin cytokine)
  Other Names: bempegaldesleukin
Drug: anti-PD-1 therapy — immunotherapy drug, monoclonal antibody
  Other Names: Pembrolizumab
Radiation: Palliative Radiation — radiation to relieve symptoms

SUMMARY:
This trial will evaluate safety and efficacy of the combination of anti-PD1, NKTR-214, and palliative radiation therapy in patients with recurrent or metastatic squamous cell carcinoma of the head and neck. Twenty-four participants will be enrolled to evaluate the efficacy of this combination.

DETAILED DESCRIPTION:
Following an informed consent process, participants will receive anti-PD-1 therapy with 200 mg of pembrolizumab and NKTR-214 at 0.006 mg/kg. Palliative radiation therapy will then be delivered to tumor sites causing or felt by the treating physician to have a high potential for causing symptoms with either 8 Gy X 3 or 4 Gy X 5 completed 3 to 7 days prior to cycle 2 of anti-PD1 and NKTR-214. Combined anti-PD-1 and NKTR-214 will then be delivered each subsequent cycle.

Efficacy will be measured by overall response rate (ORR), progression free survival (PFS), overall survival (OS), clinical benefit (CB), and duration of response with ORR the primary outcome being compared to historical control data. Toxicity will be evaluated prior to administration of each 21-day cycle, while receiving NKTR-214 followed by every four months after the participant is off trial. Health related quality of life questionnaires will be completed with cycle 1 and 2 and then every 4 cycles thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately
* Qualify for anti-PD-1 therapy based on current guidelines at the time of registration. This includes the standard requirement for the participant's tumor to have been previously determined to express PD-L1 with a combined positive score ≥ 1, as determined by an FDA-approved test.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2 within 30 days prior to enrollment
* Histologically proven diagnosis of head and neck squamous cell carcinoma that is metastatic or recurrent disease that is surgically incurable
* Prior cancer treatment other than anti-PD-1 therapy must be completed at least 30 days prior to registration and the participant must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to ≤ Grade 1 or baseline. Participants may not undergo concurrent anti-cancer treatment during treatment with protocol therapies. This includes no treatment with growth factors, tyrosine kinase inhibitors, tumor-specific antibodies, or cytotoxic chemotherapies such as cisplatin. Participants who have previously or are currently taking an anti-PD-1 therapy are eligible for this study if they meet eligibility criteria 2. Participants who have previously taken any other immune checkpoint inhibitor are eligible as long as they have completed that treatment at least 30 days prior to registration and meet all other eligibility criteria.
* Participants with central nervous system (CNS) metastases are eligible if the CNS lesions are stable for at least 2 months and if tapered off treatment doses of systemic corticosteroids for at least 2 weeks prior to enrollment on the trial. Management with maintenance physiologic doses of corticosteroids (equivalent doses of prednisone ≤ 10 mg daily) is acceptable.
* Participants must have an "index" tumor that: 1) is deemed by the treating radiation oncologist to potentially benefit from palliative radiation 2) is amenable to biopsy, 3) is ≥ 1 cm in longest dimension.
* Demonstrate adequate organ function as defined in the table below; all screening labs to be obtained within 30 days prior to enrollment

  * White blood cell (WBC) ≥ 3,000/mm3
  * Absolute Neutrophil Count (ANC) ≥ 1,500/mm3
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Platelets ≥ 100,000/mm3
  * Serum creatinine ≤ 2.0 mg/dL
  * Total Bilirubin ≤ 2.0 × upper limit of normal (ULN) (< 3.0 for subjects with Gilbert's Syndrome)
  * Aspartate aminotransferase (AST) ≤ 3 × ULN
  * Alanine aminotransferase (ALT) ≤ 3 × ULN
* Females of childbearing potential must have a negative serum pregnancy test within 14 days prior to enrollment and must agree to use effective contraception during active treatment and for 5 months after last dose of pembrolizumab and/or NKTR-214. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for ≥ 12 consecutive months.
* As determined by the enrolling physician or protocol designee, ability of the participant to understand and comply with study procedures for the entire length of the study

Exclusion Criteria:

* Subjects with significant intercurrent illnesses per physician discretion
* Subjects with active or acute infections or active peptic ulcers, unless these conditions are adequately corrected or controlled, in the opinion of the treating physician
* Subjects with a diagnosed auto-immune disease (exceptions: subjects with controlled diabetes mellitus type I, thyroid disease, rheumatoid arthritis, vitiligo and alopecia areata not requiring treatment with immunosuppressants are eligible)

  * Subjects with a history of diabetes mellitus requiring systemic therapy within the past 3 months (i.e. either oral hypoglycemic agents or insulin) must have a documented Hemoglobin A1c < 8.0 % within 90 days of registration.
* Subjects with known genetic conditions causing pre-disposition to radiotherapy (RT) toxicity (i.e.: Li-Fraumeni, ATM deficiency, active scleroderma, etc.)
* Participants with a prior diagnosis of cerebrovascular accident (CVA) or transient ischemic attack (TIA)
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study)
* Known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least three years prior to enrollment
* Prolonged Fridericia's corrected QT interval (QTcF) > 450 ms for men and > 470 ms for women at time of enrollment
* Subjects with symptoms of ischemic cardiac disease, congestive heart failure, or myocardial infarction within 6 months of registration and/or uncontrolled cardiac rhythm disturbance
* Subjects with a pulmonary embolism, deep vein thrombosis, or prior clinically significant venous or non-CVA/TIA arterial thromboembolic event (e.g., internal jugular vein thrombosis) within 3 months prior to enrollment

  * Patients with a history of a venous or arterial thromboembolic event must be asymptomatic prior to enrollment and must be receiving a stable regimen of therapeutic anticoagulation (low molecular weight heparin (LMWH) or direct oral anticoagulation (DOAC)). Use of coumadin is permitted; however, therapeutic dosing should target a specific international normalized ratio (INR) stable for at least 4 weeks prior to enrollment. NKTR-214 has the potential to down-regulate metabolizing enzymes for coumadin for approximately 1 week after administration of each dose of NKTR-214. Due to the possibility of drug-drug interactions between coumadin and NKTR-214, frequent monitoring of INR and ongoing consideration of dose adjustments are warranted throughout the patient's participation on study.
* Subjects with significant psychiatric disabilities or seizure disorders if considered unsafe in the opinion of the treating physician
* Subjects with symptomatic pleural effusions or ascites
* Subjects with organ allografts
* Subjects who require, or are likely to require, systemic treatment doses of corticosteroids, or other immunosuppressive drugs, or have used them within 2 weeks of registration (clarification: subjects receiving physiologic maintenance or replacement doses of systemic steroids or inhaled steroids are eligible)
* Subjects with known human immunodeficiency virus (HIV) infection, active or chronic hepatitis B or hepatitis C infection, or with clinical evidence of hepatitis 15. Subjects with known hypersensitivity to IL2 or those who experienced significant immune-related AEs requiring treatment with steroids or other immunosuppressant therapy during prior treatment with ipilimumab, or anti- PD-1/PD-L1 checkpoint blockade therapy 16. Subjects who cannot provide independent, legal, informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Morris, MD, PhD, Study Chair — University of Wisconsin, Madison; Paul Harari, MD, Study Chair — University of Wisconsin, Madison; Adam Burr, MD, PhD, Principal Investigator — University of Wisconsin, Madison; Justine Bruce, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were consented from August 2021 to February 2022.
Groups:
- NKTR-214, Anti-PD Therapy Plus Palliative Radiation: Cycle 1 consists of anti-PD-1 therapy (200mg) and NKTR-214 (0.006 mg/kg3 administered intravenously), followed by palliative radiation (8 Gy x 3 or 4 Gy x 5 fractions) combined with anti-PD-1 therapy and NKTR-214 in cycle 2.
  In subsequent cycles participants will receive NKTR-214 and anti-PD-1.
  NKTR-214: Bempegaldesleukin (NKTR-214) is an immunotherapeutic protein prodrug specifically designed to activate the patient's immune system for the treatment of cancer by providing a controlled, sustained signal to the interleukin-2 (IL-2) receptor pathway (pharmacological classification: immunostimulatory interleukin cytokine)
  anti-PD-1 therapy: immunotherapy drug, monoclonal antibody
  Palliative Radiation: radiation to relieve symptoms
Period: Overall Study
Arm/Group | NKTR-214, Anti-PD Therapy Plus Palliative Radiation
Started | 5
On Treatment | 5
C1D8 | 5
C2D8 | 4
C3D8 | 4
Off Treatment | 4
30 Days Post Treatment | 4
Completed | 4
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | NKTR-214, Anti-PD Therapy Plus Palliative Radiation
Number analyzed (Participants) | 5
Age, Customized [Count of Participants; unit: Participants]
  50-59 years old | 3
  60-69 years old | 1
  70-79 years old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is the percentage of participants whose cancer shrinks or disappears after treatment. ORR will include confirmed complete response (CR) + confirmed partial response (PR) and will be determined as per RECIST1.1, by investigator assessment.
Time Frame: up to 7 months (at Standard-of-care imaging 3 to 6 months after Cycle 1)
Measure: Count of Participants; unit: Participants
Arm/Group | NKTR-214, Anti-PD Therapy Plus Palliative Radiation
Number analyzed (Participants) | 5
Participants | 2

2. Secondary Outcome: Number of Participants With Adverse Events Greater Than or Equal to Grade 3
Description: Toxicities ≥ Grade 3 is defined by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Toxicities not "unrelated" to treatment, will be considered treatment-related. Adverse events are evaluated by the physician graded from 1-5 where 1 = mild, 2 = moderate, 3 = severe, 4 = life threatening, and 5 = death.
Time Frame: up to 14 months (study terminated early)
Measure: Count of Participants; unit: Participants
Arm/Group | NKTR-214, Anti-PD Therapy Plus Palliative Radiation
Number analyzed (Participants) | 5
Participants | 2

3. Secondary Outcome: Summary of Adverse Events Greater Than or Equal to Grade 3 by Count of Participants Who Experienced Them
Description: Toxicities ≥ Grade 3 is defined by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Toxicities not "unrelated" to treatment, will be considered treatment-related. Adverse events are evaluated by the physician and graded from 1-5 where 1 = mild, 2 = moderate, 3 = severe, 4 = life threatening, and 5 = death.
Time Frame: up to 14 months (study terminated early)
Measure: Count of Participants; unit: Participants
Groups:
- Grade 3: Total Grade 3 Adverse Events Among 5 Patients Evaluable for Toxicity
- Grade 4: Total Grade 4 Adverse Events Among 5 Patients Evaluable for Toxicity
- Grade 5: Total Grade 5 Adverse Events Among 5 Patients Evaluable for Toxicity
Arm/Group | Grade 3 | Grade 4 | Grade 5
Number analyzed (Participants) | 5 | 5 | 5
Participants
  Weight Loss | 1 | 0 | 0
  Dry Mouth | 1 | 0 | 0
  Sepsis | 0 | 0 | 1
  Skin Ulceration | 1 | 0 | 0
  Thrush | 1 | 0 | 0
  Lymphocyte Count Decreased | 0 | 1 | 0
  Hyperthyroidism | 1 | 0 | 0
  Hypoalbuminemia | 1 | 0 | 0
  Hyponatremia | 0 | 1 | 0
  Hypercalcemia | 0 | 1 | 0

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is the average length of time after the start of treatment in which a person is alive, and their cancer does not grow or spread. PFS is defined as the time from day 1 of treatment until the criteria for disease progression is met as defined by RECIST1.1 or death as a result of any cause.
Time Frame: up to 14 months (study terminated early)
Measure: Median (Standard Deviation); unit: months
Arm/Group | NKTR-214, Anti-PD Therapy Plus Palliative Radiation
Number analyzed (Participants) | 5
months | 4.2 (4.1)

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from day 1 of treatment until death as a result of any cause.
Time Frame: up to 14 months (study terminated early)
Measure: Mean (Standard Deviation); unit: months
Arm/Group | NKTR-214, Anti-PD Therapy Plus Palliative Radiation
Number analyzed (Participants) | 5
months | 13.6 (9.3)

6. Secondary Outcome: Number of Participants With Clinical Benefit (CB)
Description: CB will include confirmed complete response (CR) + confirmed partial response (PR) + stable disease at ≥ 6 months (SD) and will be determined as per RECIST1.1.
Time Frame: up to 14 months (study terminated early)
Measure: Count of Participants; unit: Participants
Arm/Group | NKTR-214, Anti-PD Therapy Plus Palliative Radiation
Number analyzed (Participants) | 5
Participants | 2

7. Secondary Outcome: Duration of Response
Description: Duration of response is the period measured from the time that measurement criteria are met for complete or partial response (whichever status is recorded first) until the date that recurrent or progressive disease is objectively documented.
Time Frame: up to 14 months (study terminated early)
Measure: Mean (Standard Deviation); unit: months
Arm/Group | NKTR-214, Anti-PD Therapy Plus Palliative Radiation
Number analyzed (Participants) | 5
months | 6.59 (3.7)

8. Secondary Outcome: Health Related Quality of Life as Measured by EORTC QLQ-C30: Global and Functional Sub-Scores
Description: European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) is a measure of health-related quality of life for cancer patients participating in clinical trials. It scores the following domains from 0-100 where higher global or functional scores indicate increased quality of life and higher symptom scores indicate increased symptoms: Global health status (QL2), Physical functioning (PF2), Role functioning (RF2), Emotional functioning (EF), Cognitive functioning (CF), and Social functioning (SF).
Time Frame: Baseline at screening, cycle (C)1 day (D)8 (about 2 weeks on study), C2D8 (about 5 weeks on study), C3D8 (about 8 weeks on study), 30-day post (about 12 weeks on study)
Measure: Median (Standard Deviation); unit: score on a scale
Groups:
- NKTR-214, Anti-PD Therapy Plus Palliative Radiation (Screening): EORTC QLQ-C30: Global and Functional Sub-Scores prior to treatment
- NKTR-214, Anti-PD Therapy Plus Palliative Radiation (C1D8): Cycle 1 consists of anti-PD-1 therapy (200mg) and NKTR-214 (0.006 mg/kg3 administered intravenously), followed by palliative radiation (8 Gy x 3 or 4 Gy x 5 fractions) combined with anti-PD-1 therapy and NKTR-214 in cycle 2.
- NKTR-214, Anti-PD Therapy Plus Palliative Radiation (C2D8); NKTR-214, Anti-PD Therapy Plus Palliative Radiation (C3D8): Participants will receive NKTR-214 and anti-PD-1. Palliative Radiation: radiation to relieve symptoms.
- NKTR-214, Anti-PD Therapy Plus Palliative Radiation (30-day Post): EORTC QLQ-C30: Global and Functional Sub-Scores Post Treatment
Arm/Group | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (Screening) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (C1D8) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (C2D8) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (C3D8) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (30-day Post)
Number analyzed (Participants) | 5 | 5 | 4 | 4 | 4
score on a scale
  QL2 | 66.7 (34.56) | 50.0 (22.82) | 70.8 (20.83) | 75.0 (40.82) | 62.5 (29.27)
  PF2 | 100 (29.81) | 93.3 (28.05) | 90.0 (11.55) | 93.3 (7.70) | 93.3 (7.70)
  RF2 | 100.0 (44.72) | 100.0 (22.36) | 66.7 (16.67) | 91.7 (15.96) | 83.3 (19.25)
  EF | 66.7 (25.00) | 66.7 (20.07) | 87.5 (17.18) | 83.3 (21.92) | 83.3 (21.92)
  CF | 83.3 (13.94) | 83.3 (21.73) | 100.0 (0) | 91.7 (15.96) | 83.3 (25.00)
  SF | 83.3 (13.9) | 83.3 (20.41) | 100.0 (25.00) | 91.7 (31.55) | 91.7 (23.57)

9. Secondary Outcome: Health Related Quality of Life as Measured by EORTC QLQ-C30: Symptom Sub-Scores
Description: European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) is a measure of health-related quality of life for cancer patients participating in clinical trials. It scores the following domains from 0-100 where higher symptom scores indicate increased symptoms: Fatigue (FA), Nausea and vomiting (NV), Pain (PA), Dyspnea (DY), Insomnia (SL), Appetite loss (AP), Constipation (CO), Diarrhea (DI), Financial difficulties (FI)
Time Frame: as for outcome 8
Measure: Median (Standard Deviation); unit: score on a scale
Groups:
- NKTR-214, Anti-PD Therapy Plus Palliative Radiation (Screening): EORTC QLQ-C30: Symptom Sub-Scores prior to treatment
- NKTR-214, Anti-PD Therapy Plus Palliative Radiation (30-day Post): EORTC QLQ-C30: Symptom Sub-Scores Post Treatment
Arm/Group | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (Screening) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (C1D8) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (C2D8) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (C3D8) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (30-day Post)
Number analyzed (Participants) | 5 | 5 | 4 | 4 | 4
score on a scale
  FA | 13.3 (20.76) | 20.0 (10.11) | 16.7 (9.43) | 13.3 (17.53) | 23.3 (18.36)
  NV | 0.0 (21.73) | 16.7 (19.00) | 16.7 (20.97) | 16.7 (25.00) | 0.0 (16.67)
  PA | 33.3 (40.14) | 33.3 (21.73) | 25.0 (21.52) | 25.0 (28.87) | 16.7 (39.38)
  DY | 0.0 (14.91) | 0.0 (18.26) | 0.0 (16.67) | 0.0 (16.67) | 0.0 (16.67)
  SL | 33.3 (27.89) | 33.3 (27.89) | 16.7 (31.91) | 16.7 (47.14) | 0.0 (33.33)
  AP | 33.3 (40.82) | 33.3 (33.33) | 16.7 (31.91) | 16.7 (31.91) | 0.0 (50.00)
  CO | 0.0 (18.26) | 0.0 (43.46) | 0.0 (33.33) | 0.0 (16.67) | 0.0 (16.67)
  DI | 0.0 (0) | 0.0 (0) | 0.0 (16.67) | 0.0 (16.67) | 16.7 (19.25)
  FI | 0.0 (43.46) | 0.0 (29.81) | 0.0 (16.67) | 0.0 (16.67) | 0.0 (16.67)

10. Secondary Outcome: Health Related Quality of Life as Measured by EORTC QLQ-H&N35 Sub-Scores
Description: European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire - Head and Neck (EORTC QLQ-H&N35) is comprised of the following subscales, scored from 0-100 where higher scores indicate increased symptoms: Pain (HNPA), Swallowing (HNSW), Senses problem (HNSE), Speech problems (HNSP), Trouble with social eating (HNSO), Trouble with social contact (HNSC), Less sexuality (HNSX), Teeth (HNTE), Opening mouth (HNOM), Dry mouth (HNDR), Sticky saliva (HNSS), Coughing (HNCO), Felt ill (HNFI), pain killers (HNPK), Nutritional supplements (HNNU), Feeding tube (HNFE), Weight loss (HNFL), Weight gain (HNWG)
Time Frame: as for outcome 8
Measure: Median (Standard Deviation); unit: score on a scale
Groups:
- NKTR-214, Anti-PD Therapy Plus Palliative Radiation (Screening): EORTC QLQ-H&N35 Sub-Scores prior to treatment
- NKTR-214, Anti-PD Therapy Plus Palliative Radiation (30 Days Post): EORTC QLQ-H&N35 Sub-Scores Post Treatment
Arm/Group | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (Screening) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (C1D8) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (C2D8) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (C3D8) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (30 Days Post)
Number analyzed (Participants) | 5 | 5 | 4 | 4 | 4
score on a scale
  HNPA | 25 (19.00) | 33.33 (18.26) | 20.83 (22.95) | 0 (29.17) | 29.17 (42.22)
  HNSW | 8.33 (12.63) | 8.33 (18.07) | 20.83 (27.64) | 8.33 (27.53) | 20.83 (39.89)
  HNSE | 16.67 (21.73) | 0 (36.13) | 0 (25.00) | 8.33 (31.55) | 16.67 (25.00)
  HNSP | 11.11 (14.49) | 0 (21.29) | 16.67 (19.25) | 5.56 (15.71) | 22.22 (25.66)
  HNSO | 25 (24.58) | 16.67 (36.13) | 16.67 (35.60) | 12.5 (39.31) | 45.83 (55.43)
  HNSC | 0 (12.99) | 0 (21.29) | 6.67 (22.03) | 6.67 (28.48) | 10 (28.24)
  HNSX | 0 (54.77) | 16.67 (41.83) | 0 (50.00) | 16.67 (47.14) | 16.67 (47.17)
  HNTE | 0 (14.91) | 0 (29.81) | 0 (16.67) | 0 (16.67) | 16.67 (19.25)
  HNOM | 0 (18.26) | 0 (18.26) | 16.67 (19.25) | 16.67 (19.25) | 0 (50.00)
  HNDR | 66.67 (43.46) | 66.67 (27.89) | 50 (19.25) | 50 (43.03) | 33.33 (50.00)
  HNSS | 66.67 (18.26) | 33.33 (33.33) | 33.33 (16.67) | 16.67 (31.91) | 33.34 (50.00)
  HNCO | 33.33 (23.57) | 66.67 (43.46) | 3.33 (41.93) | 16.67 (31.91) | 50 (31.91)
  HNFI | 0 (14.91) | 3.33 (23.57) | 16.67 (31.91) | 16.67 (47.14) | 0 (33.33)
  HNPK | 60 (54.77) | 80 (44.72) | 75 (50.00) | 50 (57.74) | 50 (57.74)
  HNNU | 60 (54.77) | 40 (54.77) | 75 (50.00) | 50 (57.74) | 50 (0)
  HNFE | 20 (44.72) | 20 (44.72) | 0 (0) | 0 (0) | 0 (0)
  HNWL | 40 (54.77) | 20 (44.72) | 0 (0) | 0 (0) | 75 (50.00)
  HNWG | 40 (54.77) | 20 (44.72) | 25 (50) | 25 (25) | 0 (0)

11. Secondary Outcome: Health Related Quality of Life as Measured by EQ-5D Participant Counts
Description: The EQ-5D is a 5 question measure of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression plus an overall measure of health reported on a visual analog scale. Participant counts are reported for each of 5 dimensions: mobility, self-care, usual activities, pain / discomfort, anxiety / depression.
Time Frame: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- NKTR-214, Anti-PD Therapy Plus Palliative Radiation (Baseline): EQ-5D Participant Counts prior to treatment
- NKTR-214, Anti-PD Therapy Plus Palliative Radiation (30 Days Post): EQ-5D Participant Counts 30 days post treatment
Arm/Group | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (Baseline) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (C1D8) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (C2D8) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (C3D8) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (30 Days Post)
Number analyzed (Participants) | 5 | 5 | 4 | 4 | 4
Participants
  MOBILITY: No problems / No Pain / No Anxiety | 4 | 4 | 4 | 3 | 3
  MOBILITY: Slight problems / Slight pain / Slight anxiety | 0 | 1 | 0 | 1 | 1
  MOBILITY: Moderate problems / Moderate pain / Moderate anxiety | 0 | 0 | 0 | 0 | 0
  MOBILITY: Severe problems / Severe pain / Severe anxiety | 1 | 0 | 0 | 0 | 0
  MOBILITY: Unable / Extreme pain / Extreme anxiety | 0 | 0 | 0 | 0 | 0
  SELF-CARE: No problems / No Pain / No Anxiety | 4 | 4 | 4 | 4 | 4
  SELF-CARE: Slight problems / Slight pain / Slight anxiety | 1 | 1 | 0 | 0 | 0
  SELF-CARE: Moderate problems / Moderate pain / Moderate anxiety | 0 | 0 | 0 | 0 | 0
  SELF-CARE: Severe problems / Severe pain / Severe anxiety | 0 | 0 | 0 | 0 | 0
  SELF-CARE: Unable / Extreme pain / Extreme anxiety | 0 | 0 | 0 | 0 | 0
  USUAL ACTIVITIES: No problems / No Pain / No Anxiety | 4 | 3 | 3 | 4 | 4
  USUAL ACTIVITIES: Slight problems / Slight pain / Slight anxiety | 0 | 2 | 1 | 0 | 0
  USUAL ACTIVITIES: Moderate problems / Moderate pain / Moderate anxiety | 0 | 0 | 0 | 0 | 0
  USUAL ACTIVITIES: Severe problems / Severe pain / Severe anxiety | 1 | 0 | 0 | 0 | 0
  USUAL ACTIVITIES: Unable / Extreme pain / Extreme anxiety | 0 | 0 | 0 | 0 | 0
  PAIN / DISCOMFORT: No problems / No Pain / No Anxiety | 1 | 0 | 2 | 2 | 2
  PAIN / DISCOMFORT: Slight problems / Slight pain / Slight anxiety | 2 | 2 | 1 | 0 | 0
  PAIN / DISCOMFORT: Moderate problems / Moderate pain / Moderate anxiety | 2 | 3 | 1 | 1 | 1
  PAIN / DISCOMFORT: Severe problems / Severe pain / Severe anxiety | 0 | 0 | 0 | 0 | 1
  PAIN / DISCOMFORT: Unable / Extreme pain / Extreme anxiety | 0 | 0 | 0 | 1 | 0
  ANXIETY / DEPRESSION: No problems / No Pain / No Anxiety | 2 | 3 | 2 | 2 | 3
  ANXIETY / DEPRESSION: Slight problems / Slight pain / Slight anxiety | 3 | 2 | 2 | 1 | 1
  ANXIETY / DEPRESSION: Moderate problems / Moderate pain / Moderate anxiety | 0 | 0 | 0 | 1 | 0
  ANXIETY / DEPRESSION: Severe problems / Severe pain / Severe anxiety | 0 | 0 | 0 | 0 | 0
  ANXIETY / DEPRESSION: Unable / Extreme pain / Extreme anxiety | 0 | 0 | 0 | 0 | 0

12. Other Pre Specified Outcome: Expression of PD-L1 by Histology
Description: PD-L1 expression has been shown to predict response to immunotherapy regimens. If PD-L1 expression correlates with outcome, it could be used in the future to select patients who have greatest benefit from this regimen.
Time Frame: up to 3 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Levels of IFN-γ Expressing and CD122+ T Cells in Peripheral Blood Mononuclear Cells (PBMC)
Description: Evaluation of the in vivo immune response will help better define the mechanism of action of this combination therapy.
Time Frame: up to 5 years
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Diversity and Clonality of the T Cell Receptor Repertoire by Deep Sequencing of PBMC
Description: Evaluation of the in vivo immune response will help better define the mechanism of action of this combination therapy.
Time Frame: up to 5 years
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Levels of Tumor Infiltrating Lymphocytes by Histology
Description: Evaluation of the in vivo immune response will help better define the mechanism of action of this combination therapy.
Time Frame: up to 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 14 months (study terminated early per Sponsor)
Arm/Group | NKTR-214, Anti-PD Therapy Plus Palliative Radiation
All-Cause Mortality (participants affected / at risk) | 1/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (N=5)
Sepsis (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 1
Hyponatremia (Renal and urinary disorders) | 1
Hypercalcemia (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NKTR-214, Anti-PD Therapy Plus Palliative Radiation (N=5)
Fever (General disorders) | 1
Fatigue (General disorders) | 2
Myalgias (General disorders) | 1
Anorexia (General disorders) | 1
Weight Loss (General disorders) | 1
Dry Mouth (General disorders) | 1
Pain (General disorders) | 1
Insomnia (General disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 1
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1
Thrush (Skin and subcutaneous tissue disorders) | 1
Concentration Impairment (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Gait Disturbance (Nervous system disorders) | 1
Muscle Weakness (Nervous system disorders) | 1
Hypotension (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Hyperbilirubinemia (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 3
Eosinophilia (Blood and lymphatic system disorders) | 3
Lymphocyte Count Decrease (Blood and lymphatic system disorders) | 1
Neutrophil Count Decrease (Blood and lymphatic system disorders) | 1
Hyperglycemia (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 2
Hyperthyroidism (Endocrine disorders) | 2
Hypoalbuminemia (Endocrine disorders) | 2
Creatinine Increase (Renal and urinary disorders) | 1
Hyponatremia (Renal and urinary disorders) | 1
Hypokalemia (Renal and urinary disorders) | 1

LIMITATIONS AND CAVEATS:
Study terminated early by the sponsor

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT04936841/Prot_SAP_000.pdf